CLINICAL TRIAL: NCT01303653
Title: Endoscopic Treatment of Intestinal Fistulas and Perforations
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Oregon Clinic (Other)
Responsible Party: Lee L. Swanstrom, MD, The Oregon Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LEG 1280
Record Dates: First submitted 2011-02-24; First posted 2011-02-25 (Estimated); Last update posted 2011-02-28 (Estimated); Status verified 2010-07

CONDITIONS: Gastrointestinal Fistula; Gastrointestinal Perforation
Keywords: endoscopic tissue closure,; gastro-gastric fistulas,; gastrointestinal perforations
MeSH Terms: conditions — Digestive System Fistula

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: endoscopic closure of gastrointestinal fistulas and perforations — novel endoscopic tissue closure devices will be used for endoscopic closure of gastrointestinal fistulas or perforations
  Other Names: Either the Tissue Apposition System (Ethicon Endosurgery); or the Overstitch (Apollo Endosurgery); will be used within this study for tissue closure

SUMMARY:
Gastrointestinal leaks or perforations are currently treated through either open or laparoscopic surgical procedures. The purpose of this research is to determine whether new endoscopic tools are safe and effective in the treatment of such conditions and can overcome the need of invasive surgical procedures.

DETAILED DESCRIPTION:
Novel endoscopic devices have the potential to overcome the need for invasive surgery for the treatment of gastrointestinal fistulas or perforations.

Instead of a large abdominal incision or multiple incisions with the related postoperative morbidity endoscopic techniques will be used used which require no postoperative limitation of activities. Using novel tissue closure devices, such as a Tissue Apposition System or an endoscopic suturing system, we will evaluate the potential benefit, risks and impact on the patient's quality of life of this modified surgical technique in patients having either chronic gastrointestinal fistulas or acute perforations.

ELIGIBILITY:
Inclusion Criteria:

* Gastrointestinal fistula and perforation
* Ability to undergo general anesthesia
* Ability to give informed consent

Exclusion Criteria:

* Contraindicated for esophagogastroduodenoscopy (EGD)
* Contraindicated for colonoscopy
* BMI ≥ 40
* Presence of esophageal stricture
* Altered gastric anatomy
* Intraabdominal abscess or severe inflammation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2010-10; Primary Completion 2010-10 (Estimated)

PRIMARY OUTCOMES:
Number of participants with adverse events as a measure of safety and tolerability | 6 months
  elective endoscopy to evaluate tissue closure

CONTACTS AND LOCATIONS:
Locations (1):
- Good Samaritan Hospital, Legacy Health System, Portland, Oregon, United States